CLINICAL TRIAL: NCT02260271
Title: Florida Neonatal Neurologic Network
Acronym: FN3
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201501109
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood, urine and buccal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Database Entry/Biospecimen Collection: Medical information of infants born with HIE entered into RedCap database. In addition, Blood, urine, buccal samples will be collected.
  Interventions: Other: Database Entry/Biospecimen Collection

INTERVENTIONS:
Other: Database Entry/Biospecimen Collection — blood, urine, buccal samples and medical data collected

SUMMARY:
Create a database with selected medical information on infants born with hypoxic-ischemic encephalopathy (HIE). In addition, the following samples will be collected in a bio-repository for future studies: blood, urine, and buccal samples.

DETAILED DESCRIPTION:
The purpose of this study is to create a detailed medical and sample database of infants born with HIE. Both the medical information and the samples are de-identified. Any future studies performed with the data and samples will receive Institutional Review Board (IRB) approval.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age greater than or equal to 35 weeks gestation
* Birth weight greater than or equal to 1.8 kg
* Less than or equal to 6 hours since insult occurred
* Severe hypoxic-ischemic encepholopathy (HIE)

Exclusion Criteria:

* Presence of lethal chromosomal abnormalities
* Severe IUGR
* Significant intracranial hemorrhage with a large intracranial hemorrhage (Grade III or intraparenchymal echodensity (Grade IV))

Ages: 1 Day to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants diagnosed with hypoxic-ischemic encepholopathy (HIE) at birth
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-09-09 (Actual); Primary Completion 2045-12 (Estimated); Study Completion 2045-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of blood-based biomarkers of neonatal Hypoxic Ischemic Encephalopathy (HIE) | 2 years
  Measure HIE biomarker levels in blood samples obtained in infants born with HIE.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Weiss, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided